CLINICAL TRIAL: NCT04862013
Title: Return to Sports After ACLR (RTSACL)
Brief Title: Return to Sports After ACLR
Acronym: RTSACL
Status: Completed | Type: Observational
Sponsor: crossklinik AG (Other)
Collaborators: University of Basel (Other); Basel Academy for Quality and Research in Medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: RTSACL
Record Dates: First submitted 2021-03-02; First posted 2021-04-27 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2022-07

CONDITIONS: Anterior Cruciate Ligament Injuries; Reconstruction
Keywords: anterior cruciate ligament injuries; return to sport
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients who were surgically treated with ACL reconstruction at a single clinic between 2013 and 2018 will be approached by a questionnaire regarding their return to sport after surgery. Questions will focus on the timepoint of the return, subsequent injuries, and the impact of the initial injury on the life of the patients. In addition, existing clinical data from the baseline visit and from the follow-up visits offered routinely to the patient will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* ACL injury
* surgically treated with ACL reconstruction at the crossklinik or affiliated institutions between 1.1.2013 and 31.12.2018

Exclusion Criteria:

* different treatment approach to the injury (e.g. conservative, stimulation of healing response, surgical treatment for re-rupture etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients of age ≥18, who had an ACL injury and were surgically treated with ACL reconstruction at the crossklinik or affiliated institutions between 1.1.2013 and 31.12.2018 by a small group of experienced surgeons will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Time until return to sport | All patients will be asked in a cross sectional assessment, i.e. at one specific date (planned: May 31, 2021). The distance of this time point to the time of surgery will vary between 2 and 8 years.
  This will be based on a self reporting by the patient.
Occurrence of a subsequent injury after return to sport | All patients will be asked in a cross sectional assessment, i.e. at one specific date (planned: May 31, 2021). The distance of this time point to the time of surgery will vary between 2 and 8 years.
  This will be based on the self reporting by the patient

SECONDARY OUTCOMES:
Average Muscle Strength | At 1 year follow up.
  Muscle strength is assessed by considering the flexion/extension ratio. This data will be collected retrospectively form the medical records,
Relative frequency of coping strategies | All patients will be asked in a cross sectional assessment, i.e. at one specific date (planned: May 31, 2021). The distance of this time point to the time of surgery will vary between 2 and 8 years.
  A series of questions about the impact of the injury on the life of the patients will be answered by the patients

CONTACTS AND LOCATIONS:
Locations (1):
- crossklinik AG, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
The data will be made available on request.